CLINICAL TRIAL: NCT06263608
Title: STAROSA Trial - Structured Testing and Treatment for Obstructive Sleep Apnea in Patients With Atrial Fibrillation
Brief Title: Structured Testing and Treatment for Obstructive Sleep Apnea in Patients With Atrial Fibrillation
Acronym: STAROSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Jessa Hospital (Other); Hasselt University (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUN B3002023000204
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea
Keywords: Atrial fibrillation; Obstructive sleep apnea; Cardiorespiratory polygraphy; Continuous positive airway pressure; Mobile health technology
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive | interventions — Polysomnography; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Symptomatic AF patients (Other): Eligible participants will use the NOX T3s polygraphy device for one night at home. If they have a positive obstructive sleep apnea diagnosis, they will be referred to a polysomnography examination, and subsequently treatment. Participants will also receive 3 to 6 months of semi-continuous heart rhythm monitoring with the Fitbit smartwatch (depending on whether they get treatment after obstructive sleep apnea diagnosis via polysomnography).
  Interventions: Device: (Cardio)Respiratory polygraphy (NOX T3s); Diagnostic Test: Polysomnography; Device: Devices to deliver Continuous Positive Airway Pressure (CPAP), Bilevel Positive Airway Pressure (BiPAP) or Adaptive support ventilation (ASV); Device: Fitbit smartwatch

INTERVENTIONS:
Device: (Cardio)Respiratory polygraphy (NOX T3s) — This home-based device enables the detection of obstructive sleep apnea by calculating the apnea hypopnea index (AHI).
Diagnostic Test: Polysomnography — Polysomnography allows both sleep and respiration monitoring during an overnight stay in a dedicated sleep clinic.
Device: Devices to deliver Continuous Positive Airway Pressure (CPAP), Bilevel Positive Airway Pressure (BiPAP) or Adaptive support ventilation (ASV) — Devices can be used to deliver CPAP, BiPAP, or ASV treatment to open up the airways, making breathing during sleep possible.
Device: Fitbit smartwatch — The smartwatch enables the semi-continuous monitoring of the heart rhythm via the installed FibriCheck algorithm.

SUMMARY:
The main goal of this prospective pre-post implementation study is to investigate how a structured testing and treatment program for obstructive sleep apnea using the NOX T3s device and a Fitbit smartwatch with the FibriCheck algorithm impacts the proportion of atrial fibrillation (AF) in an AF population.

Participants will wear the NOX T3s respiratory polygraphy device for one night at home. In case of a positive obstructive sleep apnea diagnosis, patients will be referred to the sleep clinic for a polysomnography examination. Patients positively diagnosed with polygraph will be monitored semi-continuously with the Fitbit smartwatch for three months. After the polysomnography examination, the positively diagnosed patients will be monitored semi-continuously for another three months after initiation of treatment (mostly continuous positive airway pressure (CPAP) treatment). Additionally, patients will be administered satisfaction, symptom burden and alcohol consumption questionnaires twice: right after the polysomnography examination and after the 3-month treatment.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most prevalent arrhythmia globally. Research has shown that AF is associated with various risk factors such as hypertension, diabetes, obesity, and obstructive sleep apnea. Obstructive sleep apnea is a sleep-disordered breathing condition that is highly prevalent in AF patients, contributing to the development and progression of AF.

Despite the high prevalence of obstructive sleep apnea in AF patients (about 62%), it often goes underrecognized and underdiagnosed. Lack of symptom reporting and easily accessible screening tools and strategies contribute to this underdiagnosis. The standard diagnostic method is through polysomnography, which, while effective, has drawbacks such as high costs, labor intensity, and time-consuming nature, making it challenging to use as a screening tool. (Cardio)respiratory polygraphy devices, such as the NOX-T3s, are gaining interest for obstructive sleep apnea detection due to their user-friendly nature, comfort, convenience, and home useability. A previous validation study showed that the NOX-T3s polygraphy device had high accuracy, sensitivity, and specificity and was also the most user-friendly for obstructive sleep apnea detection in AF patients.

Besides the screening, retrospective research has shown that obstructive sleep apnea treatment with the gold standard method, continuous positive airway pressure (CPAP), positively influences AF recurrence through improved antiarrhythmic therapy. Current literature suggests early obstructive sleep apnea diagnosis, followed by early CPAP treatment, could reduce AF recurrence. However, prospective studies supporting this are lacking. Therefore, additional information on the heart rhythm of AF patients, monitored in a (semi)-continuous manner before and after treatment initiation, would be valuable to investigate if treatment (mostly CPAP) leads to a reduction in AF events.

However, implementing a care pathway using the NOX T3s for structured obstructive sleep apnea testing and the Fitbit Versa smartwatch with the FibriCheck algorithm for the follow-up of AF recurrence in standard clinical care in an AF population still needs to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom AF (paroxysmal or persistent) is diagnosed with a 12-lead ECG
* Patients who experience symptoms of their AF (mEHRA ≥ 2a)
* Older than 18 years
* Owning a smartphone compatible with Fitbit and FibriCheck applications (i.e. recent versions of Apple iOS or Android drivers)
* Ability to sign the informed consent

Exclusion Criteria:

* Patients diagnosed with permanent AF or only atrial flutter
* Prior/recent polysomnography evaluation
* Prior/active CPAP/BiPAP/ASV treatment
* Cognitive impairment
* Inability to speak or fully understand Dutch
* Pacemaker-dependent heart rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
AF burden before and after CPAP treatment | During the entire duration of the study (2 periods of 3 months)
  The AF burden will be measured via semi-continuous FibriCheck measurements via a Fitbit smartwatch.

SECONDARY OUTCOMES:
Obstructive sleep apnea severity agreement between polygraphy and polysomnography | Result known after polysomnography examination, on average 6 weeks after the polysomnography examination
  The obstructive sleep apnea severity agreement between the NOX T3s polygraphy device and the in-hospital polysomnography examination will be assessed by evaluating AHI values.
False positive rate of polygraphy | Result known after polysomnography examination, on average 6 weeks after the polysomnography examination
  The false positive rate will be calculated using a polygraphy apnea-hypopnea index value for referral to the sleep clinic compared to polysomnography
Total sleep apnea burden | On average 3 months after initiation of obstructive sleep apnea treatment
  The total sleep apnea burden will be measured by the CPAP/BiPAP/ASV device
CPAP/BiPAP/ASV compliance | On average 3 months after initiation of obstructive sleep apnea treatment
  CPAP/BiPAP/ASV compliance will be read out from the device.
Sleep score | 3 months after first and after second period of semi-continuous monitoring with Fitbit smartwatch
  The sleep score will be determined based on Fitbit data. The score is based on sleep duration, sleep quality, and restoration. The minimum value is 0 and the maximum value is 100. The higher the value, the better the overall sleep efficiency.
Patients' AF-related symptom burden, assessed by the Leuven ARrhythmia Questionnaire (LARQ) | Right after the polysomnography examination and 3 months after obstructive sleep apnea treatment
  The Leuven ARrhythmia Questionnaire (LARQ) will be used to assess the AF symptom profile based on six symptoms: palpitations, dyspnea, chest pain, syncope, dizziness, and fatigue. The minimum score is 0 and maximum score is 100. The higher the score, the more pronounced the symptom burden.(LARQ) before and after treatment.
Patients' obstructive sleep apnea-related symptom burden, assessed by the Berlin Questionnaire (BQ) | Right after the polysomnography examination and 3 months after obstructive sleep apnea treatment
  The Berlin Questionnaire (BQ) will be used to assess the risk of sleep apnea focusing on 3 OSA symptoms (snoring, daytime sleepiness, and obesity/hypertension). For the first two symptoms, the category is positive if 2 points or more are given. The last category is positive if the patient has obesity and/or hypertension.
Patients' obstructive sleep apnea-related symptom burden, assessed by the Epworth Sleepiness Scale (ESS) | Right after the polysomnography examination and 3 months after obstructive sleep apnea treatment
  The Epworth Sleepiness Scale (ESS) will be used to assess the overall daytime sleepiness in eight situations. Minimum score is 0 and the maximum score is 24. The higher the score, the higher the chance for daytime sleepiness.
Polygraphy negative patients | 24 hours after the one-time use of the polygraphy device
  The number of polygraphy-negative patients in a general AF population will be calculated.
Patients' alcohol consumption assessed by the Alcohol Use Disorder Identification Test-Consumption (AUDIT-C) supplemented with four additional questions related to alcohol consumption | Right after the polysomnography examination and 3 months after obstructive sleep apnea treatment
  This questionnaire on alcohol consumption includes the Alcohol Use Disorder Identification Test-Consumption (AUDIT-C) supplemented with four additional questions related to alcohol consumption. The AUDIT-C consists of three questions, which can help identify who may have an active alcohol use disorder. It is scored on a scale of 0 to 12 points, with 0 points indicating no alcohol use in the past year. A higher AUDIT-C score suggests a greater likelihood of adverse effects on the individual's health and safety. The four additional questions inquire about the weekly consumption of alcohol-containing drinks, the type of drinks, their effects on sleep, and their impact on AF symptoms.

OTHER OUTCOMES:
User-friendliness of the NOX T3s polygraphy device | Right after using the polygraphy device
  The patient reported experience measure questionnaire assesses the user-friendliness and patient satisfaction of the NOX T3s PG device. The minimum score is 0, the maximum score is 40. The higher the score, the more user-friendly the device.
User-friendliness of the Fitbit-based FibriCheck monitoring | Right after the first and second period of 3 months of semi-continuous monitoring with the Fitbit smartwatch
  The patient reported experience measure questionnaire assesses the user-friendliness and patient satisfaction of the Fitbit smartwatch with FibriCheck monitoring. The minimum score is 0, the maximum score is 60. Additionally, patients are questioned about the type and long-term time of monitoring with FibriCheck.
Uptake rate of the advice to patients to undergo a polysomnography examination | Immediately after the polysomnography examination
  The uptake rate will be evaluated by assessing the number of scheduled polysomnography examination in patients with a positive polygraphy test.
Protocol adherence to smartphone heart rhythm measurements | After the first and second period of 3 months of FibriCheck monitoring with the smartphone
  The FibriCheck report will be used to evaluate whether patients were adherent to performing at least 2 spot-check measurements daily.
The quality of the FibriCheck measurements | After the first and second period of 3 months of FibriCheck monitoring with the smartphone
  The algorithm indicates low quality measurements. The number of low quality measurements will be evaluated during the follow-up compared to the good quality measurements.
Number of technical issues | During study completion after 6months of follow-up
  A troubleshooting document will be set up in which solutions will be recorded in the case of technical difficulties regarding the used devices.

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbuchel, MD, PhD, Principal Investigator — University Hospital of Antwerp
Locations (2):
- Belgium (2):
  - University Hospital of Antwerp, Edegem
  - Jessa Hospital, Hasselt

IPD SHARING:
Plan to Share IPD: No